CLINICAL TRIAL: NCT06470295
Title: On the Regulation of Hepatic Glucose Metabolism During Insulin-induced Hypoglycemia
Brief Title: Effect of C-peptide on Hypoglycemic Counterregulation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jason Winnick, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-0236
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hypoglycemia; Type 1 Diabetes
Keywords: glucagon; hepatic glucose production; C-peptide
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Sodium Chloride; C-Peptide

STUDY DESIGN:
Intervention Model Description: Each subject will undergo two metabolic studies, one where they receive an IV infusion of C-peptide during insulin-induced hypoglycemia, and one where they will receive an IV infusion of saline instead.
Who Masked: Participant, Investigator
Masking Description: During participation in these studies, the subject and the researchers will not know which treatment (C-peptide versus saline) was administered to the subject on what day until after that subject has completed the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Control- Saline (Placebo Comparator): Saline will be infused in healthy control subjects during insulin-induced hypoglycemia
  Interventions: Other: Saline
- Healthy Control- C-peptide (Active Comparator): C-peptide will be infused in healthy control subjects during insulin-induced hypoglycemia
  Interventions: Biological: C-peptide
- T1D- Saline (Placebo Comparator): Saline will be infused in T1D subjects during insulin-induced hypoglycemia
  Interventions: Other: Saline
- T1D- C-peptide (Active Comparator): C-peptide will be infused in T1D subjects during insulin-induced hypoglycemia
  Interventions: Biological: C-peptide

INTERVENTIONS:
Other: Saline — Normal saline will be infused during insulin-induced hypoglycemia
  Arms: Healthy Control- Saline; T1D- Saline
Biological: C-peptide — C-peptide will be infused during insulin-induced hypoglycemia
  Arms: Healthy Control- C-peptide; T1D- C-peptide

SUMMARY:
Iatrogenic hypoglycemia is the most prominent barrier to the safe, effective management of blood sugar in people with type 1 diabetes due to periodic over-insulinization. During insulin-induced hypoglycemia, glucagon secretion is diminished in type 1 diabetes which, in turn, reduces hepatic glucose production and increases the depth and duration of hypoglycemic episodes. We have observed that the naturally occurring protein C-peptide increases glucagon secretion in dogs during insulin-induced hypoglycemia, which increases hepatic glucose production; the experiments in this application will shed light on the translation of this finding to the human.

DETAILED DESCRIPTION:
Iatrogenic hypoglycemia is recognized as a primary barrier to the safe, effective management of blood glucose in people with type 1 diabetes (T1D). In previous experiments in the dog, we observed that C-peptide infusion augmented glucagon secretion and hepatic glucose production during insulin-induced hypoglycemia. The proposed experiments will determine the translational impact of this finding in patients with and without T1D.

Specific Aim #1 is to determine, in healthy control subjects, the effect of C-peptide co-infusion with insulin on endogenous glucose production (EGP) and counterregulatory hormone levels during hypoglycemia. This will be addressed by studying a single group of healthy subjects two times. In both studies, hypoglycemia will be induced with an intravenous (IV) infusion of insulin. During one study, C-peptide will be infused during the hypoglycemic period, and in the other study, saline will be infused. EGP is our primary variable, with secondary analyses including counterregulatory hormones and metabolic substrates.

Specific Aim #2 is to determine, in T1D patients, the effect of C-peptide co-infusion with insulin on EGP and counterregulatory hormone levels during hypoglycemia. The research plan for this Aim is very similar to that of Aim #1, with the main exception being that we will study T1D patients instead of healthy controls (e.g., two hypoglycemic clamp studies where C-peptide is administered during one study and saline during the other). In addition, the glycemic levels of these T1D patients will be monitored for 10 days prior to this visit to ensure that they do not experience hypoglycemia which could confound the data for the metabolic studies. Similar to Aim #1, EGP is our primary outcome variable, with secondary analyses including hormone and substrate levels.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 30 kg/m2

Exclusion Criteria:

* pregnant or lactating women cigarette smoking presence of HIV or hepatitis presence of cardiovascular disease presence of microvascular disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Glucagon | During procedure, up to 2.5 hours
  from plasma

SECONDARY OUTCOMES:
Hepatic glucose production | During procedure, up to 2.5 hours
  from plasma
Liver glycogen | Prior to insulin-induced hypoglycemia
  from MRS measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jason Winnick, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warner SO, Dai Y, Sheanon N, Yao MV, Cason RL, Arbabi S, Patel SB, Lindquist D, Winnick JJ. Short-term fasting lowers glucagon levels under euglycemic and hypoglycemic conditions in healthy humans. JCI Insight. 2023 Jun 22;8(12):e169789. doi: 10.1172/jci.insight.169789. PMID 37166980
- See also: Link to published paper — https://pubmed.ncbi.nlm.nih.gov/37166980/